CLINICAL TRIAL: NCT01969695
Title: An Extension Study of Venetoclax in Subjects With Advanced Non-Hodgkin's Lymphoma
Brief Title: An Extension Study of ABT-199 in Subjects With Advanced Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-835
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: ABT-199; Cancer; GDC-0199; non-Hodgkin's lymphoma; Relapsed; Refractory; Safety
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms; Recurrence | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABT-199 (Experimental): ABT-199 monotherapy
  Interventions: Drug: ABT-199

INTERVENTIONS:
Drug: ABT-199 — ABT-199 continuous once daily dosing
  Other Names: GDC-0199

SUMMARY:
This is a Phase 1, open-label, multicenter, extension study. Subjects with non-Hodgkin's lymphoma (NHL) (excluding chronic lymphocytic lymphoma [CLL], small lymphocytic lymphoma [SLL], and mantle cell lymphoma [MCL]) who completed a prior ABT-199 study, or were active and assigned to ABT-199 when the study was completed, may roll over into this extension study. Subjects will receive ABT-199 during this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed a prior ABT-199 study (and had met the criteria for a diagnosis of NHL and all other eligibility criteria for the previous study) and the investigator believes that treatment with ABT-199 is in the best interest of the subject.

Exclusion Criteria:

* Subject discontinued ABT-199 administration before completing the prior study (due to disease progression, toxicity, withdrawn consent, other).
* Subject has any medical condition that in the opinion of the investigator places the subject at an unacceptably high risk for toxicities.
* Subject has not recovered to ≤ Grade 2 clinically significant adverse effect(s)/toxicity(ies) of previous therapy.
* Subject has been diagnosed with Post-Transplant Lymphoproliferative Disease (PTLD), Burkitt's lymphoma, Burkitt-like lymphoma, lymphoblastic lymphoma/leukemia, chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), or mantle cell lymphoma (MCL).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Change in cardiac assessment findings | Measured from Day 1 up to 6 years after the last subject has enrolled in the study
  Electrocardiogram and Multi Gated Acquisition Scan and/or Echocardiogram
Percentage of subjects with adverse events | Measured up to 6 years after the last subject has enrolled in the study
  Subjects will be monitored for clinical and laboratory evidence of adverse events throughout the study
Change in clinical laboratory test results | Measured from Day 1 up to 6 years after the last subject has enrolled in the study
  Chemistry, coagulation, hematology, lymphocyte enumeration, paraproteins, urinalysis, and, if appropriate, viral polymerase chain reaction and viral serologies
Number of subjects with adverse events | Measured up to 6 years after the last subject has enrolled in the study
  Subjects will be monitored for clinical and laboratory evidence of adverse events throughout the study
Change in physical exam finding, including vital signs | Measured from Day 1 up to 6 years after the last subject has enrolled in the study
  Body temperature, weight, blood pressure, heart rate

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (3):
- United States (3):
  - University of Arizona Arthritis Center /ID# 101359, Tucson, Arizona
  - Dartmouth-Hitchcock Med Ctr /ID# 92596, Lebanon, New Hampshire
  - Hackensack Univ Med Ctr /ID# 101417, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No